CLINICAL TRIAL: NCT02512042
Title: A Multicentre, Double Blind, Active Controlled, Parallel Group, Two Arm, Bioequivalence Study With Clinical Endpoint Comparing Brinzolamide 1% Ophthalmic Suspension (Manufactured by Indoco Remedies Ltd. for Watson Pharma Pvt Ltd.), to Brinzolamide (Azopt®) 1% Ophthalmic Suspension of Alcon Laboratories, Inc., In the Treatment of Chronic Open Angle Glaucoma or Ocular Hypertension in Both Eyes
Brief Title: Bioequivalence Study With Clinical Endpoint Comparing Brinzolamide 1% Ophthalmic Suspension to Azopt® 1% Ophthalmic Suspension In the Treatment of Chronic Open Angle Glaucoma or Ocular Hypertension in Both Eyes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: WAT/BNZL/2014
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Results first posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brinzolamide 1% Ophthalmic suspension (Experimental): Brinzolamide Pharmaceutical dosage form: Ophthalmic suspension Strength: 1% Manufactured by: Indoco Remedies, Ltd for Watson Pharma Pvt. Ltd
  Interventions: Drug: Test-Brinzolamide 1% Ophthalmic suspension
- Azopt® 1% Ophthalmic suspension (Active Comparator): Azopt® (Contains Brinzolamide) Pharmaceutical dosage form: Ophthalmic suspension Strength: 1% Manufactured by: Alcon Laboratories, Inc
  Interventions: Drug: Reference-Brinzolamide 1% Ophthalmic suspension

INTERVENTIONS:
Drug: Test-Brinzolamide 1% Ophthalmic suspension
  Arms: Brinzolamide 1% Ophthalmic suspension
Drug: Reference-Brinzolamide 1% Ophthalmic suspension
  Arms: Azopt® 1% Ophthalmic suspension

SUMMARY:
This is a randomized, double blind, two-arm, parallel group, active controlled bioequivalence study, at multiple clinical trial sites designed to demonstrate bioequivalence of Brinzolamide 1% ophthalmic suspension (manufactured by Indoco Remedies Ltd. for Watson Pharma Pvt Ltd.), to Brinzolamide (Azopt®) 1% ophthalmic suspension of Alcon Laboratories, Inc. in the treatment of chronic open angle glaucoma or ocular hypertension in both eyes.

DETAILED DESCRIPTION:
Study will be conducted in adult subjects, above 18 years inclusive, males and non pregnant females, diagnosed with chronic open angle glaucoma or ocular hypertension in both eyes. Qualifying Intra Ocular Pressure (IOPs) following wash-out, at baseline (Day 0/hour 0 i.e., 8:00 am) should be ≥ 22 milli meter mercury (mm Hg) and ≤ 34 mm Hg in each eye and any asymmetry of IOP between the eyes no greater than 5 mm Hg.

Each study subject will use one drop of test or reference Ophthalmic Suspension in both the eyes three times daily at approximately 8:00am, 04:00 pm and 10:00 pm for 42 days (6 weeks). The dose and mode of treatment chosen in this study is the dosage approved by United States Food and Drug administration (US FDA) for use in treatment of patients of Chronic Open Angle Glaucoma.

The study subjects will undergo clinical evaluations throughout the study in order to assess efficacy and safety. Study subject primary endpoint evaluation will be assessed after 2 weeks (14 days) and 6 weeks (42 days) of treatment for each study subject deemed eligible for evaluation, (i.e., at Visit III - Day 14 ± 2 days and Visit IV - Day 42 ± 3 days).

The primary bioequivalence comparison is between the test and reference products for the mean difference in intraocular pressure (IOP) of both eyes at four time points, i.e., at approximately 8:00 am and 10:00 am at the Day 14 (± 2 days) and Day 42 (± 3 days) visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant females aged 18 years and above with a Body Mass Index (BMI) of 18.5 to 35 Kg/m2, with chronic open angle glaucoma or ocular hypertension in both eyes on stable ocular hypotensive treatment regimen.
2. Subjects requiring treatment of both eyes and are able to discontinue use of all ocular hypotensive medication(s) or switch ocular hypotensive medications and undergo appropriate washout period.
3. Adequate wash-out period prior to baseline of any ocular hypotensive medication. In order to minimize potential risk to subjects due to IOP elevations during the washout period, investigator may choose to substitute a parasympathomimetic or carbonic anhydrase inhibitor in place of a sympathomimetic, alpha-agonist, beta-adrenergic blocking agent, or prostaglandins. However, subjects must have discontinued all ocular hypotensive medication for the minimum washout period.
4. Baseline (Day 0/hour 0) IOP ≥ 22 mm Hg and ≤ 34 mm Hg in each eye and any asymmetry of IOP between the eyes no greater than 5 mm Hg.
5. Baseline best corrected visual acuity equivalent to 20/200 or better in each eye.
6. Study subjects must have provided IRB approved written informed consent using the latest version of the IRB informed consent form. In addition, study subjects must sign a Health Insurance Portability and Accountability Act (HIPAA) authorization, if applicable.
7. Study subjects should be literate and willing to complete the subject diary regularly as directed.
8. Study subjects must be in good health and free from any clinically significant disease apart from indication under study.
9. Females of child bearing potential (WOCBP*) must not be pregnant or lactating at baseline visit (as documented by a negative serum pregnancy test with a minimum sensitivity of 25 IU/L or equivalent units of beta-human chorionic gonadotropin (Beta-HCG) at screening and urine pregnancy at baseline.

   *All female subjects will be considered to be of childbearing potential unless they are postmenopausal. Female subjects of childbearing potential (WOCBP) are defined as sexually mature women without prior hysterectomy, or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for the past 12 or more months are still considered to be of childbearing potential, if the amenorrhea is possibly due to other causes, including prior chemotherapy, anti-estrogens, or ovarian suppression. Postmenopausal women (defined as women who have been amenorrheic for at least 12 consecutive months, in the appropriate age group, without other known or suspected primary cause) or women who have been sterilized surgically or who are otherwise proven sterile (i.e., total hysterectomy, or bilateral oophorectomy with surgery at least 4 weeks prior to randomization) are not considered WOCBP. Subjects who have undergone tubal ligation are NOT considered as surgically sterile.
10. Female subjects of childbearing potential must be willing to use an acceptable form of birth control from the day of the first dose administration to 30 days after the last administration of IP. For the purpose of this study the following are considered acceptable methods of birth control: oral or injectable contraceptives, contraceptive patches, Depo-Provera® (Medroxyprogesterone acetate- stabilized for at least 3 months); vaginal contraceptive; contraceptive implant; double barrier methods (e.g. condom and spermicide); Nuvaring vaginal hormonal birth control, IUD, or abstinence with a second method of birth control should the subject become sexually active. A sterile sexual partner is NOT considered an adequate form of birth control.
11. All male subjects must agree to use accepted methods of birth control with their partners, from the day of the first dose administration (to 30 days after the last administration of study drug). Please see acceptable forms for "Female" birth control above. Abstinence is an acceptable method of birth control for males.
12. Study subjects must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required scheduled study visits.
13. Study subjects must be willing to refrain from using any other treatments for Chronic Open Angle Glaucoma (COAG), other than the investigational product.

Exclusion Criteria:

1. Females who are pregnant, breast feeding, or planning a pregnancy during the course of the study and for 30 days after last study dose.
2. Females of childbearing potential who do not agree to utilize an adequate form of contraception.
3. Current or past history of severe hepatic or renal impairment.
4. Current or history within two months prior to baseline of significant ocular disease, e.g., corneal edema, uveitis, ocular infection, or ocular trauma in either eye.
5. Current corneal abnormalities that would prevent accurate IOP readings with the Goldmann applanation tonometer e.g. corneal dystrophy, corneal abrasions, corneal ulcers, keratitis, keratoconus and keratoglobus.
6. Functionally significant visual field loss
7. Contraindication to brinzolamide or sulfonamide therapy or known hypersensitivity to any component of brinzolamide or sulfonamide therapy
8. Use at any time prior to baseline of intraocular corticosteroid implant.
9. Use within one week prior to baseline of contact lens
10. Use within two weeks prior to baseline of: 1) topical ophthalmic corticosteroid, or 2) topical corticosteroid
11. Use within one month prior to baseline of: 1) systemic corticosteroid or 2) high-dose salicylate therapy defined as 325mg taken on three consecutive days.
12. Use within six months prior to baseline of intravitreal or subtenon injection of ophthalmic corticosteroid
13. Underwent within six months prior to baseline any other intraocular surgery (e.g., cataract surgery)
14. Underwent within twelve months prior to baseline: refractive surgery, filtering surgery or laser surgery for IOP reduction
15. Amblyopia - only one sighted eye
16. Severe retinal disease or other severe ocular pathology, such as glaucomatous damage with a cup/disc ratio greater than 0.8, split fixation, or functionally significant (in the investigators' opinion) visual field loss
17. History or presence of significant alcoholism or drug abuse in the past one year
18. History or presence of significant smoking (more than 20 cigarettes or any other equivalent tobacco product/day)
19. History of hematologic disorders other than mild anemia
20. Severe, unstable, or uncontrolled cardiovascular or pulmonary disease
21. Systolic blood pressure less than 90 mm Hg or more than 140 mm Hg, Diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg and Pulse rate less than 50 beats/minute or more than 100 beats/minute
22. Any form of glaucoma other than chronic open-angle glaucoma
23. Therapy with an investigational agent within the past 30 days
24. Clinically significant hematologic and / or biochemical abnormalities based on laboratory testing
25. Subjects who are in the investigator's best judgment at risk of visual field or visual acuity worsening as a consequence of participation of trial.
26. Chronic use of any systemic medication that may affect IOP with less than three month stable dosing regimen (i.e., sympathomimetic agents, beta-adrenergic blocking agents, alpha agonists, alpha-adrenergic blocking agents, calcium channel blockers, angiotensin -converting enzyme inhibitors, etc.)
27. Use of any prescribed medication during last two weeks or Over the Counter (OTC) medicinal products during the last one week preceding the first dosing that is affecting the IOP or result in drug-drug interaction with the study drug.
28. Major illness, as per investigator discretion, during 3 months before screening
29. Subjects who are employees of site or Clinical research organization (CRO) or sponsor or immediate family of employees
30. Participating in a clinical study within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 973 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - David Wirta, MD, Newport Beach, California
  - Shettle Eye Research, Inc., Largo, Florida
  - AMB Research Center, Inc., Miami, Florida
  - Eye Care Centers Management, Inc., Morrow, Georgia
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Heart of America Eye Care PA, Shawnee Mission, Kansas
  - Ophthalmology Associates, St Louis, Missouri
  - Las Vegas Physicians Research Group, Henderson, Nevada
  - Keystone Research Ltd., Austin, Texas
  - Keystone Research Ltd., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The populations for this study included the Randomized Population, Safety Population and Per Protocol Population.
Groups:
- Generic Brinzolamide Ophthalmic Suspension USP 1%; Azopt® (Brinzolomide Ophthalmic Suspension USP 1%): Study subjects used one drop in both eyes three times daily for 42 days.
Period: Overall Study
Arm/Group | Generic Brinzolamide Ophthalmic Suspension USP 1% | Azopt® (Brinzolomide Ophthalmic Suspension USP 1%)
Started | 495 | 478
Completed | 472 | 453
Not Completed | 23 | 25
Not completed — Adverse Event | 0 | 4
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Non-compliance with study drug | 1 | 2
Not completed — Lost to Follow-up | 5 | 2
Not completed — Other | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Generic Brinzolamide 1% Ophthalmic Suspension; Azopt® 1% Ophthalmic Suspension: Study subjects used one drop in both eyes three times daily for 42 days.
- Total: Total of all reporting groups
Arm/Group | Generic Brinzolamide 1% Ophthalmic Suspension | Azopt® 1% Ophthalmic Suspension | Total
Number analyzed (Participants) | 495 | 478 | 973
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (14.50) | 53.0 (14.19) | 52.9 (14.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 206 | 428
  Male | 273 | 272 | 545
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 20 | 36
  Not Hispanic or Latino | 431 | 417 | 848
  Unknown or Not Reported | 48 | 41 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 414 | 402 | 816
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 13 | 27
  White | 67 | 61 | 128
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Iris Colour [Count of Participants; unit: Participants]
  Blue | 18 | 16 | 34
  Green | 7 | 7 | 14
  Grey | 21 | 31 | 52
  Hazel | 15 | 10 | 25
  Brown | 282 | 265 | 547
  Black | 152 | 149 | 301

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Intraocular Pressure (IOP) of Both Eyes Between the Two Treatment Groups at Four Time Points
Description: The primary efficacy end point is the mean difference in intraocular pressure (IOP) of both eyes between the two treatment groups at four time points, i.e., at approximately 8:00 am (hour 0; before the morning drop) and 10:00 am (hour 2; after the morning drop) at the Day 14 (week 2) and Day 42 (week 6) visits
Time Frame: Day 14 and 42 at 8AM and 10AM
Population: Participants in Per Protocol Population who met inclusion/exclusion criteria, instilled a pre-specified proportion of the scheduled doses for the specified duration of the study, who did not miss scheduled applications for more than 3 days, and completed evaluations at Day 14 and Day 42 within the visit window.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Generic Brinzolamide Ophthalmic Suspension USP 1% | Azopt® (Brinzolomide Ophthalmic Suspension USP 1%)
Number analyzed (Participants) | 489 | 475
mmHg
  8AM Visit Day 14: number analyzed (Participants) | 430 | 429
  8AM Visit Day 14 | 19.35 (2.860) | 19.75 (2.874)
  8AM Visit Day 42: number analyzed (Participants) | 432 | 416
  8AM Visit Day 42 | 18.53 (2.894) | 18.66 (2.851)
  10AM Visit Day 14: number analyzed (Participants) | 429 | 428
  10AM Visit Day 14 | 18.70 (2.805) | 19.18 (2.710)
  10AM Visit Day 42: number analyzed (Participants) | 432 | 415
  10AM Visit Day 42 | 17.94 (2.734) | 18.16 (2.824)
Statistical Analysis 1: Comparison: Generic Brinzolamide Ophthalmic Suspension USP 1% vs Azopt® (Brinzolomide Ophthalmic Suspension USP 1%); Test type: Equivalence — The limits of each two-sided 95% confidence interval of the treatment difference (test-reference) for mean IOP of both eyes at approximately 8:00 (hours 0, before the morning drop) at the Day 14 visit should be within +/-1.5mm Hg, and should be within +/-1.0mm Hg for majority of time points using the PP population; Mean Difference (Net) = -0.36, 95% CI 2-sided [-0.69 to -0.03]
Statistical Analysis 2: Comparison: Generic Brinzolamide Ophthalmic Suspension USP 1% vs Azopt® (Brinzolomide Ophthalmic Suspension USP 1%); Test type: Equivalence — The limits of each two-sided 95% confidence interval of the treatment difference (test-reference) for mean IOP of both eyes at approximately 8:00 hour on Day 42 should be within +/-1.5mm Hg, and should be within +/- 1.0mm Hg for majority of time points using the PP population; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.43 to 0.22]
Statistical Analysis 3: Comparison: Generic Brinzolamide Ophthalmic Suspension USP 1% vs Azopt® (Brinzolomide Ophthalmic Suspension USP 1%); Test type: Equivalence — The limits of each two-sided 95% confidence interval of the treatment difference (test-reference) for mean IOP of both eyes at approximately 10:00 hour on Day 14 should be within +/-1.5mm Hg, and should be within +/-1.0mm Hg for majority of time points using the PP population; Mean Difference (Net) = -0.40, 95% CI 2-sided [-0.71 to -0.09]
Statistical Analysis 4: Comparison: Generic Brinzolamide Ophthalmic Suspension USP 1% vs Azopt® (Brinzolomide Ophthalmic Suspension USP 1%); Test type: Equivalence — The limits of each two-sided 95% confidence interval of the treatment difference (test-reference) for mean IOP of both eyes at approximately 10:00 hour on Day 42 should be within +/-1.5mm Hg, and should be within +/-1.0mm Hg for majority of time points using the PP population; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.50 to 0.13]

ADVERSE EVENTS:
Time Frame: Baseline up to 45 days
Description: Adverse events were collected from participants who were randomized and received the study drug.
Arm/Group | Generic Brinzolamide 1% Ophthalmic Suspension | Azopt® 1% Ophthalmic Suspension
Serious Adverse Events (participants affected / at risk) | 0/489 | 0/475
Other Adverse Events (participants affected / at risk) | 55/489 | 57/475
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Generic Brinzolamide 1% Ophthalmic Suspension (N=489) | Azopt® 1% Ophthalmic Suspension (N=475)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Asthenopia (Eye disorders) | 1 (1) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 1 (1) | 0 (0)
Conjunctival disorder (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 5 (5) | 2 (2)
Excessive eye blinking (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 20 (21) | 7 (7)
Eye pain (Eye disorders) | 4 (4) | 5 (5)
Eye pruritus (Eye disorders) | 3 (4) | 1 (2)
Eyelid dermatochalasis (Eye disorders) | 0 (0) | 1 (1)
Eyelid irritation (Eye disorders) | 0 (0) | 1 (1)
Eyelid margin crusting (Eye disorders) | 0 (0) | 3 (3)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 3 (3) | 3 (3)
Ocular hyperaemia (Eye disorders) | 5 (6) | 3 (3)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Punctuate keratitis (Eye disorders) | 1 (2) | 1 (1)
Vision blurred (Eye disorders) | 6 (6) | 12 (14)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (2) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 3 (3)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitic (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Mycobacterium tuberculosis complex test positive (Investigations) | 0 (0) | 1 (1)
Vital dye staining cornea present (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 3 (6) | 9 (10)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.